CLINICAL TRIAL: NCT05737706
Title: A Phase 1/2 Multiple Expansion Cohort Trial of MRTX1133 in Patients With Advanced Solid Tumors Harboring a KRAS G12D Mutation
Brief Title: Study of MRTX1133 in Patients With Advanced Solid Tumors Harboring a KRAS G12D Mutation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Formulation challenges
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA246-0005; CA246-0005 (Other: Bristol-Myers Squibb Protocol ID); 1133-001 (Other: Mirati Therapeutics Protocol ID)
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor; Advanced Solid Tumor; Non-small Cell Lung Cancer; Colo-rectal Cancer; Pancreatic Adenocarcinoma
Keywords: Non-Small Cell Lung Cancer; NSCLC; colorectal cancer; CRC; PDAC; KRAS; G12D; Solid Tumor; Advanced Solid Tumor; Malignant; Pancreatic Cancer; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms | interventions — KRASG12D inhibitor MRTX1133

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1/1B (Experimental): Dose Escalation/Evaluation
  Interventions: Drug: MRTX1133
- Phase 2 (Experimental): MRTX1133 recommended Phase 2 dose administered to separate cohorts of patients with selected solid tumor malignancies with KRAS G12D mutation to include the following: NSCLC, PDAC, CRC, Other Solid Tumors
  Interventions: Drug: MRTX1133

INTERVENTIONS:
Drug: MRTX1133 — KRAS G12D Inhibitor

SUMMARY:
A Phase 1/2 study of MRTX1133 in solid tumors harboring a KRAS G12D mutation.

DETAILED DESCRIPTION:
This first-in-human clinical trial will begin with an exploration of MRTX1133 dose and regimen. As potentially viable regimens are identified, Phase 1b expansion cohorts may be implemented to ensure collection of sufficient safety and PK information, and early evidence of clinical activity are available to recommend Phase 2 regimens. In Phase 2, separate cohorts of patients by histological diagnosis and/or baseline characteristics will be evaluated for the clinical activity and efficacy of MRTX1133.

This study was terminated prior to phase 2 initiating. Only phase 1 of the study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy harboring KRAS G12D mutation in tumor tissue or ctDNA.
* Unresectable or metastatic disease.
* Patients must have received standard therapies appropriate for their tumor type and stage; first-line treatment for PDAC for certain cohorts.
* Presence of tumor lesions to be evaluated per RECIST v1.1:

  1. in the Phase 1 dose escalation cohorts, patients must have measurable or evaluable disease.
  2. in the Phase 1b and Phase 2 cohorts, patients must have measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function.
* Age ≥ 18 years

Exclusion Criteria:

* Active brain metastases or carcinomatous meningitis.
* Prior treatment with a KRAS G12D inhibitor (Phase 1b & Phase 2 only).
* History of significant hemoptysis or hemorrhage within 4 weeks of the first dose of study treatment.
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions likely to alter absorption of study treatment or result in inability to swallow oral medications.
* History of malignant small bowel obstruction.
* Cardiac abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Phase 1: Number of Patients who Experience Dose-Limiting Toxicity | 21 Days
Phase 1/1b: Number of patients who experience a treatment-related adverse event | Up to 2 years
Phase 2: Objective response rate (ORR) | 2 years
Phase 2: Duration of response (DOR) | 2 years
Phase 2: Progression free survival (PFS) | 2 years
Phase 2: Overall survival (OS) | 2 years

SECONDARY OUTCOMES:
Area under plasma concentration versus time curve (AUC) | up to 4 days
Time to achieve maximal plasma concentration (Tmax) | up to 4 days
Maximum observed plasma concentration (Cmax) | up to 4 days
Terminal elimination half-life (t1/2) | up to 4 days
Apparent total plasma clearance when dosed orally (CL/F) | up to 4 days
Apparent volume of distribution when dosed orally (Vz/F) | up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (14):
  - Local Institution - 311, Phoenix, Arizona
  - Local Institution - 309, New Haven, Connecticut
  - Local Institution - 301, Lady Lake, Florida
  - Local Institution - 306, Baltimore, Maryland
  - Local Institution - 308, Boston, Massachusetts
  - Local Institution - 310, Boston, Massachusetts
  - Local Institution - 314, Grand Rapids, Michigan
  - Local Institution - 312, New York, New York
  - Local Institution - 303, Nashville, Tennessee
  - Local Institution - 302, Houston, Texas
  - Local Institution - 304, San Antonio, Texas
  - Local Institution - 313, San Antonio, Texas
  - Local Institution - 305, Fairfax, Virginia
  - Local Institution - 307, Seattle, Washington

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com